CLINICAL TRIAL: NCT07061535
Title: Efficacy and Safety of Sintilimab Combined With Tafolecimab and Chemotherapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer (STAR-SCLC)：A Prospective, Single Arm Trial
Brief Title: Sintilimab Combined With Tafolecimab and Chemotherapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer
Acronym: STAR-SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025LSYD0847H
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC); Extensive Stage Lung Small Cell Cancer; Extensive-Stage Small-Cell Lung Cancer; Extensive Disease Small Cell Lung Cancer
Keywords: Tafolecimab; Sintilimab; immunotherapy; PCSK9 inhibitor; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — sintilimab; Etoposide; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Tafolecimab combined with Sintilimab and Chemotherapy as the first-line treatment regimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafolecimab + Sintilimab + Chemotherapy (Experimental): Eligible patients will receive 4 cycles of Tafolecimab (300 mg, sc, d1, Q3W) in combination with Sintilimab (200 mg, iv, d1, Q3W), along with etoposide and either carboplatin (AUC 5 mg/mL/min) or cisplatin (75 mg/m2) for up to 4 to 6 cycles. Subsequently, they will receive maintenance therapy with Sintilimab and Tafolecimab until disease progression, the occurrence of intolerable toxicities, or the completion of 2 years of treatment. Etoposide (100 mg/m2) will be administered intravenously on days 1, 2, and 3 of each 3-week cycle, while carboplatin or cisplatin will be given intravenously on day 1 of each 3-week cycle.
  Interventions: Drug: Tafolecimab; Drug: Sintilimab (approved); Drug: Etoposide; Drug: Carboplatin / Cisplatin

INTERVENTIONS:
Drug: Tafolecimab — Patients will receive Tafolecimab 300 mg every 3 weeks.
Drug: Sintilimab (approved) — Patients will receive Sintilimab 200 mg every 3 weeks.
Drug: Etoposide — Patients will recieve Etoposide (100 mg/m2) intravenously on days 1, 2, and 3 of each 3-week cycle.
Drug: Carboplatin / Cisplatin — Patients will receive carboplatin (AUC 5 mg/mL/min) or cisplatin (75 mg/m2) intravenously on day 1 of each 3-week cycle for up to 4 to 6 cycles.

SUMMARY:
This is a single arm, multi-center clinical trial. The goal of this clinical trial is to evaluate the efficacy, safety and biomarkers of Tafolecimab combined with Sintilimab and Chemotherapy as first-line treatment for patients with extensive-stage small cell lung cancer (ES-SCLC). Tafolecimab is a recombinant fully humanized monoclonal antibody against proprotein convertase subtilisin/kexin type 9 (PCSK-9), which can reduce low-density lipoprotein-C levels and increase the expression level of major histocompatibility complex class I (MHC-I) on tumor cells. Sintilimab is a fully humanized IgG4 monoclonal antibody targeting programmed cell death protein 1 (PD-1).

DETAILED DESCRIPTION:
Eligible patients will receive 4 cycles of Tafolecimab (300mg, sc, d1, Q3W) in combination with Sintilimab (200mg, iv, d1, Q3W), along with etoposide and either carboplatin (AUC 5 mg/mL/min) or cisplatin (75 mg/m2) administered intravenously on days 1, 2, and 3 of each 3-week cycle for up to 4 to 6 cycles. Subsequently, patients will receive maintenance therapy with Sintilimab and Tafolecimab until disease progression, the occurrence of intolerable toxicities, or the treatment duration reaches 2 years. If the investigator assesses potential evidence of clinical benefit, continuing treatment after disease progression is permitted.

PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) of Tafolecimab combined with Sintilimab and chemotherapy as first-line treatment regimens for patients with extensive-stage small cell lung cancer (ES-SCLC).

SECONDARY OBJECTIVES:

I. To evaluate the safety of of Tafolecimab combined with Sintilimab and chemotherapy as first-line treatment regimens for patients with ES-SCLC.

II. To evaluate the PFS rate, objective response rate (ORR), disease control rate (DCR), duration of response (DOR), overall survival (OS) rate and OS of Tafolecimab combined with Sintilimab and chemotherapy as first-line treatment regimens for patients with ES-SCLC.

TERTIARY OBJECTIVES:

I. To evaluate whether Tafolecimab combined with Sintilimab and chemotherapy as first-line treatment for patients with ES-SCLC could upregulate the expression of MHC-I on SCLC tumor cells.

II. To explore tissue and liquid biopsy biomarkers that may be predictive of response or primary resistance to Tafolecimab combined with Sintilimab and chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years, ECOG performance status 0-1;
* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC) according to Veterans Administration Lung Study Group criteria;
* Previously not receiving systemic treatment for ES-SCLC;
* Greater than or equal to 1 measurable lesion exists according to RECIST v1.1;
* Expected survival >= 12 weeks;
* Adequate organ system functions (no blood transfusion or component blood use within 14 days before testing).

Key Exclusion Criteria:

* Previously receiving systemic anti-tumor therapy for ES-SCLC;
* Combined SCLC (mixed SCLC and NSCLC histological types) or transformed SCLC confirmed by histological or cytological examination;
* Receiving other investigational drugs or participated in other interventional clinical studies within 4 weeks before signing the informed consent form;
* Receiving systemic immunostimulant treatment within 4 weeks before enrollment;
* Active central nervous system (CNS) metastases (asymptomatic patients with stable lesions allowed);
* Severe cardiovascular disease;
* Severe chronic/active infections requiring systemic antibacterial, antifungal or antiviral treatment within 2 weeks before enrollment;
* Active hepatitis B virus (HBV)/ hepatitis C virus (HCV)/ human immunodeficiency virus (HIV) infection;
* Active autoimmune diseases, a history of interstitial lung disease, or other uncontrolled systemic diseases;
* Pregnancy or lactation;
* Having a disease that requires systemic corticosteroids or other immunosuppressants to be treated within ≤14 days before enrollment;
* Requiring at least monthly or more frequent drainage of pleural and/or pericardial or peritoneal effusion;
* Using attenuated live vaccines, or planned to receive attenuated live vaccines within 28 days before enrollment;
* Known to be allergic to Sintilimab or Tafolecimab or its excipients, having a history of severe allergic reaction to any monoclonal antibody, or having a history of allergy to cisplatin, carboplatin or etoposide;
* Toxicity caused by previous anti-cancer treatment has not recovered to baseline or stable state at the time of enrollment;
* Creatinine clearance rate < 60 mL/min (cisplatin) or < 45 mL/min (carboplatin)
* Uncontrolled or symptomatic hypercalcemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival as Assessed by RECIST v1.1 | From enrollment to the end of treatment at 12 months
  Progression-free survival (PFS) refers to the period from the start of combined treatment until any objectively recorded tumor progression occurs or until the patient's death (for patients lost to follow-up, it is the last follow-up time; for patients still alive at the end of the study, it is the date of the follow-up termination) as assessed by RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate as Assessed by RECIST v1.1 | From enrollment to the end of treatment at 12 months
  Objective response rate (ORR) refers to the proportion of patients whose tumors have shrunk to a certain extent and maintained that state for a certain period of time, including cases of complete response (CR) and partial response (PR) as assessed by RECIST v1.1.
Progression-free Survival Rate as Assessed by RECISIT v1.1 | From enrollment to the end of treatment at 6 months and 12 months
  6-month and 12-month progression-free survival rate refers to the proportion of patients whose time from the start of treatment to any objectively recorded tumor progression or patient death is equal to or greater than 6 months and 12 months.
Overall Survival Rate as Assessed by RECISIT v1.1 | From enrollment to the end of treatment at 12 months and 24 months
  12-month and 24-month overall survival rate refers to the proportion of patients whose time from the first administration of the drug to any cause of death was greater than or equal to 12 months and 24 months.
Disease Control Rate as Assessed by RECISIT v1.1 | From enrollment to the end of treatment at 12 months
  Disease control rate refers to the proportion of patients whose tumors have shrunk to a certain extent and maintained that state for a certain period of time. It includes cases of complete response (CR), partial response (PR), and stable disease (SD).
Duration of Response as Assessed by RECISIT v1.1 | From enrollment to the end of treatment at 12 months
  Duration of response refers to the duration from the time when the patient's condition is first confirmed as response (CR or PR) until the first record of progressive disease (PD) or death due to any reason (whichever occurs first).
Percentage of Participants with Treatment-Related Adverse Events as Assessed by NCI-CTCAE v5.0 | From enrollment to the end of treatment at 12 months
Overall survival as Assessed by RECISIT v1.1 | From enrollment to the end of treatment at 24 months
  The time period from the first administration of the drug until death due to any cause (for patients who were lost to follow-up, it is the last follow-up time; for patients who were still alive at the end of the study, it is the date of the follow-up conclusion).

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Hunan Cancer Hospital/the Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Science, Jinan, Shandong
  - Department of Thoracic Medical Oncology, Zhejiang Cancer Hospital, Hangzhou Institute of Medicine (HIM), Chinese Academy of Sciences, Hangzhou, Zhejiang
  - First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zugazagoitia J, Osma H, Baena J, Ucero AC, Paz-Ares L. Facts and Hopes on Cancer Immunotherapy for Small Cell Lung Cancer. Clin Cancer Res. 2024 Jul 15;30(14):2872-2883. doi: 10.1158/1078-0432.CCR-23-1159. PMID 38630789
- [Background] Mei W, Faraj Tabrizi S, Godina C, Lovisa AF, Isaksson K, Jernstrom H, Tavazoie SF. A commonly inherited human PCSK9 germline variant drives breast cancer metastasis via LRP1 receptor. Cell. 2025 Jan 23;188(2):371-389.e28. doi: 10.1016/j.cell.2024.11.009. Epub 2024 Dec 9. PMID 39657676
- [Background] Liu X, Bao X, Hu M, Chang H, Jiao M, Cheng J, Xie L, Huang Q, Li F, Li CY. Inhibition of PCSK9 potentiates immune checkpoint therapy for cancer. Nature. 2020 Dec;588(7839):693-698. doi: 10.1038/s41586-020-2911-7. Epub 2020 Nov 11. PMID 33177715
- [Background] Ma S, He Z, Liu Y, Wang L, Yang S, Wu Y, Chen H, Wu Y, Wang Q. Sintilimab plus anlotinib as second or further-line therapy for extensive disease small cell lung cancer: a phase 2 investigator-initiated non-randomized controlled trial. EClinicalMedicine. 2024 Mar 14;70:102543. doi: 10.1016/j.eclinm.2024.102543. eCollection 2024 Apr. PMID 38516099